CLINICAL TRIAL: NCT03540602
Title: Polyphenol Rich Supplementation on Markers of Recovery From Intense Resistance Exercise
Acronym: PRSRE
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Jacksonville University (Other)
Collaborators: Specnova, inc (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: Polyphenol Supplementation
Record Dates: First submitted 2018-02-26; First posted 2018-05-30 (Actual); Last update posted 2018-05-30 (Actual); Status verified 2018-05

CONDITIONS: Muscle Soreness
Keywords: Polyphenol rich supplementation; Tart cherry; Lifting; Recovery
MeSH Terms: conditions — Myalgia

STUDY DESIGN:
Intervention Model Description: 20 male participants will start with a familiarization visit where they will receive either the placebo supplement or the polyphenol rich supplement that they will take for 7 days. After taking the supplement, the participants will come back and run through the acute resistance exercise protocol as well as return the next day for a post test. Next, the participants will undergo a "wash out" phase where they will not take any supplementation. At the end of these 2 weeks, the participants will then take the other supplement (i.e. if they took the polyphenol rich supplement in the first phase they will take the placebo supplement in the second phase). After a week of taking their assigned supplement, participants will complete the acute resistance exercise protocol and the post test.
Who Masked: Participant, Investigator
Masking Description: To ensure that all subjects and researchers are unaware of the treatment assignments we will have one outside individual that will possess the knowledge of which subjects are given which supplement and which were given a placebo. This information will remain confidential until the study has been concluded. At the conclusion of the study, participants will be informed of which condition they were assigned. in an event of an emergency or the participant decides not to participate his condition will be revealed.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator): Rice flour capsule
  Interventions: Other: Placebo Oral Capsule [CEBOCAP]
- Polyphenol Rich Supplement (Active Comparator): NordicCherry Tart Cherry Extract Powder 500 mg in capsule form
  Interventions: Dietary Supplement: Tart Cherry

INTERVENTIONS:
Dietary Supplement: Tart Cherry — NordicCherry Tart Cherry Extract Powder 500 mg from Specnova, inc
  Other Names: NordicCherry Tart Cherry Extract Powder 500 mg
  Arms: Polyphenol Rich Supplement
Other: Placebo Oral Capsule [CEBOCAP] — Rice flour
  Arms: Placebo

SUMMARY:
Strength training is commonly used as an intervention to increase muscle mass, thus improving a person's ability to undertake activities of daily living, or enhance athletic performance. The strength training regimen itself, while ultimately having beneficial effects, causes muscle fibers to be damaged, which the body has to recover from. As the body recovers, it rebuilds the muscle tissue and after multiple consecutive bouts of strength training, the muscle eventually becomes larger and stronger. Thus, it is the recovery from strength training exercise that ultimately determines how well the body adapts. Where inadequate recovery could eventually lead to overtraining and/or injury, optimizing the recovery process from strength training could maximize strength training adaptations. This concept of optimizing recovery has led to development of many supplements, including antioxidants, which may reduce the damage associated with strength training activities and therefore enhance positive adaptations. The purpose of this study is to assess the ability of a polyphenol rich supplementation to aid the recovery process from a demanding bout of resistance exercise

ELIGIBILITY:
Inclusion Criteria:

* 6 months of resistance training experience with barbel back squat exercise

Exclusion Criteria:

* Not currently taking any antioxidant supplements, not currently using any hormone replacement therapy or anabolic androgenic steroids.

Ages: 21 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Must be male
Enrollment: 20 (Estimated)
Dates: Start 2018-05-01 (Actual); Primary Completion 2018-08 (Estimated); Study Completion 2018-08 (Estimated)

PRIMARY OUTCOMES:
Assessment of Oxidative Stress | 7 weeks
  Blood analyses will be used, 8 mL of blood will be taken from the participant six times per condition. The blood will be centrifuged to separate the serum/ plasma and analyzed by enzyme- linked immunosorbent assay (ELISA) for c- reactive protein and creatine kinase, and oxidative damage

SECONDARY OUTCOMES:
Muscle soreness | 7 weeks
  Subjects will mark a line on a 10cm scale that corresponds to the amount of muscular soreness they currently perceive
Vertical Jump Performance | 7 weeks
  Subjects will be instructed to stand on a NeuroCom Balance Manager forceplate with hands on hips. Subjects will then be instructed to perform 3 consecutive vertical jumps, as high as possible with minimal time between jumps. The jumps will later be assessed for power production.

CONTACTS AND LOCATIONS:
Overall Officials: Heather Hausenblaus, Principal Investigator — Jacksonville University
Locations (1):
- Jacksonville University, Jacksonville, Florida, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Reid MB. Invited Review: redox modulation of skeletal muscle contraction: what we know and what we don't. J Appl Physiol (1985). 2001 Feb;90(2):724-31. doi: 10.1152/jappl.2001.90.2.724. PMID 11160074
- [Result] Alessio HM, Goldfarb AH, Cutler RG. MDA content increases in fast- and slow-twitch skeletal muscle with intensity of exercise in a rat. Am J Physiol. 1988 Dec;255(6 Pt 1):C874-7. doi: 10.1152/ajpcell.1988.255.6.C874. PMID 3202155
- [Result] Blair SN, Cheng Y, Holder JS. Is physical activity or physical fitness more important in defining health benefits? Med Sci Sports Exerc. 2001 Jun;33(6 Suppl):S379-99; discussion S419-20. doi: 10.1097/00005768-200106001-00007. PMID 11427763
- [Result] Powers SK, Jackson MJ. Exercise-induced oxidative stress: cellular mechanisms and impact on muscle force production. Physiol Rev. 2008 Oct;88(4):1243-76. doi: 10.1152/physrev.00031.2007. PMID 18923182